CLINICAL TRIAL: NCT00905151
Title: Evaluation of the Performance of GFR Estimating Equations in HIV Positive Patients
Brief Title: HIV and Kidney Function Study
Status: Completed | Type: Observational
Sponsor: Tufts Medical Center (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); University of Alabama at Birmingham (Other); University of Minnesota (Other); Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB # 8761
Record Dates: First submitted 2009-05-15; First posted 2009-05-20 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-02

CONDITIONS: HIV Infections; AIDS
Keywords: HIV positive; AIDS; antiretroviral; Kidney disease; Antiretroviral Therapy
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; HIV Seropositivity; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Whole and urine will be retained for future testing.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV Positive: Across-sectional analysis of 200 HIV+ patients with varying levels of kidney function

SUMMARY:
Current methods to assess kidney function have not been tested in people who have HIV/AIDS population. Given effects of the disease as well as potential effects of the medications, it is possible that the methods currently used to assess kidney function are not accurate. This purpose of this study is to evaluate methods to assess kidney function the HIV population. The investigators hypothesize that tenofovir causes a decrease in the secretion of creatinine which would cause an elevation in blood levels without affecting actual glomerular filtration rate (GFR).

DETAILED DESCRIPTION:
General description: The overall study procedure requires assessment of eligibility and safety for inclusion in the study (through a "screening questionnaire" and "health screening visit") and if eligible, a one day study visit ("Study visit").

Screening questionnaire All subjects, whether they are interviewed during a clinic visit or call in response to fliers, will be give the pre-screening questionnaire. This will be given to people who voluntarily express interest in the study. Participants who do not disclose any conditions that would exclude them from participating will be invited to a health screening visit.

Health screening visit The purpose of the pre-study health screening is to perform a more detailed assessment than is provided in the screening questionnaire to determine if potential subjects are eligible to participate in the study. A member of the research team will first read the consent form with the subject, describe the health screening and study visits, and answer any questions that the subject has regarding the nature of the study and/or study procedures. The screening visit will consist of the following:

* Reading and signing the study consent. The subject will be given a copy of the consent.
* Collection of information on demographics and current and past health history.
* Ascertain participants medical history through participant interview and a review of his/her medical record
* A physical exam, which will include measuring and recording vital signs (temperature, blood pressure, heart rate, breathing rate), height, weight (if not documented in medical record in past 3 months).
* Collection of a blood sample for laboratory testing, if required, as described in Table 4.
* Pre-menopausal women of child-bearing potential we will undergo a serum pregnancy test, using a small amount of blood from the sample collected above.
* Ascertainment of current and recent past medications.

If the subject is a patient at Tufts Medical Center, a research team member may access the potential participant's medical record after the subject has signed the consent form to further screen for potential exclusion criteria, ascertain laboratory test results that are necessary for determining eligibility, and confirm the medical history provided by the potential participant and medication list. If the participant is not a patient at Tufts Medical Center, then the research team member will obtain permission to obtain the participant's medical record from his/her physician.

For non-pregnant women of childbearing age (pre-menopausal) who are sexually active, use of an acceptable birth control method will be required for participation. They will be requested to sign a statement of compliance prior to participating in the study stating that they are employing one of the below-listed forms of contraception between the screening and study visits.

* condoms with spermicide
* diaphragm with spermicide
* injectable contraceptives (Depoprovera)
* transdermal contraceptives (Ortho-Evra and Nuvaring)
* intrauterine device (IUD)
* permanent sterilization (i.e. tubal ligation, vasectomy, Essure)
* abstinence from sexual activity
* hysterectomy
* oral contraceptives

If the study visit occurs 1 week or more after the health screening, the female subjects will undergo a second, urine-based pregnancy test on the morning of the study visit. Given the small dose of iohexol administered during the study visit, which is rapidly filtered by the kidneys, continued use of birth control following the completion of the study visit will not be required.

If a potential subject is taking trimethoprim containing medications or cimetidine., the study physician will discuss with the attending physician whether it is safe for the person to stop these medications for one week prior to the study. If not, then the person will be excluded from participation. If a potential subject is taking non-steroidal anti-inflammatory agents or medications that block the renin-angiotension system, the study physician will discuss with the potential participant and the attending physician whether maintenance of stable dose of these medications is possible. If a change in the subject's medication regimen is required immediately prior to the study visit, the subject will be rescheduled for a later date.

Eligibility will be determined by the principal investigator or other physician co-investigators based on the medical history obtained from the participant, and their medical records and the results of the laboratory test that were included in the medical record or obtained during the health screening visit). Eligible subjects will be contacted to see if they remain interested in participating in the study. A study visit date will then be scheduled. All subjects will receive a stipend for the health screening (see Section G.8).

Preparation for a study visit: A urine jug and a detailed set of instructions for completing the 24 hour urine collection will be mailed to the subject.

Subjects taking medications that interfere with creatinine whose physicians approved temporary discontinuation of the medication will be reminded by a phone call from the study coordinator to stop these medications 1 week prior to the study visit at this time. Subjects will also be asked not to take any multivitamins or calcium supplements on the day of the study as undigested tablet may interfere with the quality of the DEXA scan.

A research team member will contact the subject by telephone 2-3 days before the visit to ensure that the subject fully understands the instructions for completing the urine collection and has ceased taking medications that interfere with creatinine. The research team member will request that subjects with diabetes to bring all medications, administration devices (e.g. insulin syringes or controlled delivery devices), and their personal blood sugar monitoring devices (i.e. glucometers) with them on the day of the study visit.

A research team member will order the iohexol from the pharmacy.

Study visit: Non-diabetic subjects will be requested to fast overnight and to avoid changes in non-steroidal anti-inflammatory agents or medications that block the renin-angiotension system. Subjects with diabetes will be asked to eat a light breakfast the morning of the study visit. Subjects will be asked to maintain adequate oral hydration and to ingest two to three glasses of non-caffeinated beverages prior to arrival on the morning of the study visit to facilitate a timed urine collection during the study visit. If the subject feels that he/she is unable to void upon arrival, he/she will be given 2 to 3 additional non-caffeinated beverages and will be given approximately 1 beverage every hour for the remainder of the study visit.

The 24 hour urine that was collected the previous day by the participant will be given to the research team member upon arrival for the study. If the participant forgets to collect then 24 h urine or is in the midst of the collection, then the intra-study timed urine collection will be utilized for the analysis. If the participant has forgotten the container at home, arrangements will be made to collect the container within the next 2 days.

The nursing staff will measure and record the subject's height, weight, blood pressure, temperature, pulse rate, respiration rate, confirm that the subject has not experienced any changes in physical/psychological health since the screening.

The timed urine collection will begin when the participant first has the urge to void. The nursing staff will record the time of the first void and the participant will be asked to collect all urine voided during the remainder of the study visit in a collection container. To facilitate complete bladder emptying, the participant will be given a glass (approximately 6 ounces) of a non-caffeinated beverage every hour until the end of the study visit. As outlined above, if three weeks or more has elapsed since the health screening, women of childbearing age will be administered a urine pregnancy test using an aliquot of the intra-study timed urine collection. Subjects with diabetes will be asked to check their blood sugar with their own equipment or the nursing staff at the CTRC will use the CTRC's equipment. The study physician will be informed of low or high blood sugars.

A saline lock and/or intravenous line will be inserted at two different sites and a baseline blood and a separate sample for tissue banking (10 mL, optional) will be collected. After taking the baseline blood, 5 mL of iohexol(Omnipaque 300; 300 mg/mL of organic iodine) will be administered by a nurse at the Clinical and Translational Research Center (CTRC) over a period of approximately 15 seconds through an IV port, followed by a flush with approximately 10 mL of 0.9% normal saline solution. This intravenous line through which the iohexol was administered will then be removed. The syringe will be weighted to the nearest tenth gram on the same scale before and after injection. Blood samples for plasma clearance measurements will be obtained from the second IV line, which will remain in place throughout the course of the study visit. To maintain the patency of the IV access, normal saline will be administered at a rate of approximately 20-30 c.c. per hour from a 500 c.c. bag of normal saline.

The administration of iohexol will be considered time 0. Following the iohexol administration, blood samples will be taken at approximately 10, 30, 120, and 240 minutes from the second intravenous line. For participants with estimated GFR less than 45 ml/min per 1.73 m2, as determined from the screening visit or the subject's medical record, a sample will be drawn at 360 minutes. The exact time of the sample will be recorded.

After the 30 minute blood sample, participants will be fed a breakfast consisting of a standardized protein content. They will also receive a lunch of similar protein content. Subjects with diabetes will be given a meal that is consistent with their treatment regimen. Subjects will be asked to administer their medications and check their blood sugar levels during the course of the study visit as they would normally do, in the manner prescribed by their treating physician. If the subject is at the CTRC past 6 PM, he/she will also receive dinner.

The Dual-Energy X-ray Absorptiometry (DEXA) scan may be scheduled prior to the start of the GFR measurement or following the entire GFR visit if timing is best for the participant and the DEXA scan. It may be performed on a separate day. Prior to the scan, subjects will be asked to remove any metal objects (e.g. belts, earrings, jewelry, etc). Subjects may be requested to void prior to initiating the scan. During the scan, subjects will be asked to lie flat on the table for approximately 5-10 minutes while the scan takes place.

Participants are free to move around during the GFR test. At the conclusion of the GFR test, the second intravenous line will be removed. Subjects will remain at the CTRC for at least 30 minutes following removal of the IV line. During that time, nursing staff will re-measure and record the subject's vital signs (height, weight, blood pressure, temperature, pulse rate, respiration rate). The participants will be asked to void prior to leaving the CTRC to ensure complete urine collection over the study visit. The nurse will record the stop time of the urine collection. Upon successful completion of a study visit, subjects will receive a stipend.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older
* Confirmed HIV positive status
* Treatment with stable antiretroviral medications for a period of at least 3 months prior to the study

Exclusion Criteria:

* Persons less than 18 years of age. Children are excluded due to the fact that they are still growing. Growth causes levels of creatinine to change differently than in adults, thus requiring the use of age-specific GFR estimating equations.
* Women who are either pregnant or who intend to become pregnant during the period of time in which the study visits will occur.
* Allergy to any of the contrast media used or a known allergy to iodine or shellfish. Subjects who are not sure if they have an iodine allergy because they have not eaten shellfish nor have never received contrast dye will be excluded from participation.
* Inability to cease taking medications that affect creatinine levels (e.g. trimethoprim containing medications, cimetidine) for one week prior to the study visit
* Inability to maintain stable regimen of non-steroidal anti-inflammatory agents, angiotension converting enzyme inhibitors and or angiotension receptor blockers for one week prior to study visit.
* Women who are breastfeeding
* Current treatment with amiodarone
* Current treatment with metformin
* Acute exacerbation of asthma or chronic obstructive lung disease in the past three months requiring hospitalization or oral steroid therapy
* Inadequate venous access
* People with kidney failure (currently undergoing or having received peritoneal dialysis or hemodialysis treatment within the past three months or estimated GFR (eGFR) < 15 ml/min per 1.73 m2)
* End stage conditions such as cirrhosis
* Active treatment for cancer
* Progressive neurological diseases
* Severe gastric immotility
* History of cognitive or physical impairments that will not allow completion of the study
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from hospital based practices as well as from the community.
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2009-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lesley A Stevens, MS MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
N/A, this study was not funded by the NIH

REFERENCES:
- [Background] Okparavero AA, Tighiouart H, Krishnasami Z, Wyatt CM, Graham H, Hellinger J, Inker LA. Use of glomerular filtration rate estimating equations for drug dosing in HIV-positive patients. Antivir Ther. 2013;18(6):793-802. doi: 10.3851/IMP2676. Epub 2013 Aug 20. PMID 23963249
- [Result] Inker LA, Wyatt C, Creamer R, Hellinger J, Hotta M, Leppo M, Levey AS, Okparavero A, Graham H, Savage K, Schmid CH, Tighiouart H, Wallach F, Krishnasami Z. Performance of creatinine and cystatin C GFR estimating equations in an HIV-positive population on antiretrovirals. J Acquir Immune Defic Syndr. 2012 Nov 1;61(3):302-9. doi: 10.1097/QAI.0b013e31826a6c4f. PMID 22842844

RESULTS

PARTICIPANT FLOW:
Groups:
- HIV Positive: A cross-sectional analysis of 200 HIV+ patients with varying levels of kidney function
Period: Overall Study
Arm/Group | HIV Positive
Started | 206
Completed | 200
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | HIV Positive
Number analyzed (Participants) | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 194
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 145

OUTCOME MEASURES:

1. Primary Outcome: Performance of Glomerular Filtration Rate (GFR) Estimating Equations
Description: Overall bias, median difference (95% confidence interval), mL/min per 1.73 m^2, assessed as the median difference between the measured and estimated GFR across all estimated GFR levels, with positive values indicating an underestimation of measured GFR.
Time Frame: Blood samples for plasma iohexol clearance were taken at approximately 10, 30, 120, and 240 minutes post-iohexol dose.
Measure: Median (95% Confidence Interval); unit: mL/min per 1.73 m^2
Arm/Group | HIV Positive
Number analyzed (Participants) | 200
mL/min per 1.73 m^2
  MDRD study | 10.9 [8.0 to 14.0]
  CKD-EPI creatinine | 5.4 [2.7 to 7.9]
  CKD-EPI cystatin C | 4.3 [1.2 to 7.7]
  CKD-EPI creatinin-cystatin | 6.4 [3.1 to 9.3]

ADVERSE EVENTS:
Arm/Group | HIV Positive
Serious Adverse Events (participants affected / at risk) | 0/206
Other Adverse Events (participants affected / at risk) | 0/206

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No